CLINICAL TRIAL: NCT03427216
Title: A Randomized Double Blind Placebo Controlled Cross-over Trial of Baclofen and Diazepam Suppositories for the Management of Pelvic Floor Myalgia
Brief Title: Baclofen/Diazepam Supps for Treatment of Pelvic Floor Myalgia
Acronym: BDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. John A. Thiel Medical Professional Corporation (Other)
Responsible Party: Principal Investigator, John Thiel, Clinical Professor, Dr. John A. Thiel Medical Professional Corporation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Jthiel
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Pelvic Floor Dyssynergia
MeSH Terms: interventions — Baclofen; Diazepam; Suppositories

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Baclofen/diazepam supp (Active Comparator): Insert vaginal suppository once daily
  Interventions: Drug: Baclofen/diazepam
- Vaginal Placebo supp (Placebo Comparator): Insert vaginal suppository once daily
  Interventions: Drug: Vaginal placebo

INTERVENTIONS:
Drug: Baclofen/diazepam — Vaginal suppository placed once daily, patients will record pelvic pain daily on a VAS scale, sexual satisfaction and quality of life on a standardized questionnaire weekly
  Other Names: Lioresal
  Arms: Vaginal Baclofen/diazepam supp
Drug: Vaginal placebo — Vaginal suppository placed once daily, patient will record pelvic pain daily on a VAS scale, sexual satisfaction and quality of life on a standardized questionnaire weeky.
  Other Names: suppository
  Arms: Vaginal Placebo supp

SUMMARY:
This study is a randomized, placebo controlled double blind cross over trial. Patients presenting with pelvic floor myalgia will be asked to complete a series of standardized questionnaires to assess their pain, quality of life and sexual function and satisfaction. They will be randomized to either a treatment group or placebo group and will use the supplied suppositories once daily for 2 months. They will then undergo a one month "washout" after which they will be placed in the cross over group for a second two months of treatment.

Primary outcome measure: change in Visual Analogue Scale for Pain (VAS-P) scores before and after treatment Secondary outcome measures: change in Female Sexual Function Index (FSFI), Patient Global Impression of Improvement (PGI-I), and Short Form Health Survey (SF-12) before and after treatment

DETAILED DESCRIPTION:
Chronic pelvic pain is a complex multi-faceted problem that places a substantial burden on the healthcare resources. In Canada, the average hospital related cost for women requiring surgery or inpatient admission for chronic pelvic pain is $25 million each year. Chronic pelvic pain is defined as either persistent pain for at least 6 months or "recurrent episodes of abdominal/pelvic pain, hypersensitivity, or discomfort, often associated with elimination changes and sexual dysfunction in the absence of an organic etiology." Chronic pelvic pain is common and affects women of all ages and backgrounds. 15-20% of women have chronic pelvic pain lasting for more than 1 year.

Pelvic floor myalgia is an important and common contributor to chronic pelvic pain that may be present alone or may co-exist with other gynecological, urological, colorectal, and musculoskeletal medical conditions. The International Urogynecological Association/International Continence Society joint report published in February 2017 defines pelvic floor myalgia as pain in the musculature of the pelvic floor.6 Patients with high-tone pelvic floor dysfunction (HTPFD) have levator hypercontractility and present with pain with internal vaginal examination and intercourse. In a 2011 prospective cross-sectional study by Fitzgerald et al., 63% of patients with self-reported chronic pelvic pain examined by a physician and 73.7% of patients examined by a physiotherapist were found to have pelvic floor myalgia. Although pelvic floor myalgia is a common condition encountered in gynecology, it is frequently an unrecognized and under-treated component of chronic pelvic pain. Pelvic floor myalgia has a significant impact on the patient's quality of life. Persistent chronic pain may result in patient's anxiety, low mood, depression, sleep disturbances, feeling of hopelessness and helplessness, frustration, and psychological distress.

The first line of treatment for pelvic floor myalgia is pelvic floor muscle relaxation. Reducing the resting tone of pelvic floor musculature has been shown to improve chronic pelvic pain. Current treatment options for pelvic floor myalgia include pelvic floor physiotherapy, Thiele massage, biofeedback with electrical stimulation, behavioural modifications, acupuncture, medications such as antidepressants,1 trigger point injections with botulin A toxin, warm sitz baths, and neuromodulation.

Recently, intravaginal diazepam has been used an off-label treatment option for high-tone pelvic floor myalgia. Diazepam is a benzodiazepine derivative that has both antispasmotic and anxiolytic activity. It is used as a muscle relaxant and enhances the inhibitory action of gamma-amino butyric acid (GABA) on neuronal excitability, resulting in decreased action potentials. The benefit of local therapy is the avoidance of the common side effects of benzodiazepines such as drowsiness, fatigue, and ataxia. Currently, evidence is lacking in regards to the effectiveness of intravaginal diazepam on treatment of chronic pelvic pain. The 2010 retrospective chart review of 26 patients by Rogalski et al. revealed clinically significant reduction in Visual Analogue Scale for Pain (VAS-P) and Female Sexual Function Index (FSFI) with diazepam suppositories used for 30 days as an adjuvant therapy to pelvic floor physiotherapy and intramuscular trigger point injections. Similarly, the 2011 study revealed 62% improvement in symptoms with intravaginal diazepam.

Baclofen is a skeletal muscle relaxant. It is a GABA-B receptor agonist which is commonly used for treating spasticity. The literature on topical baclofen use in pelvic floor dysfunction is minimal. Topical therapy is advantageous to avoid the common systemic side effects such as drowsiness, hypotonia, hypotension, and headache. A retrospective study examining the use of topical baclofen for provoked vulvodynia showed an improvement in pain and sexual function.

Baclofen may also be used in combination with diazepam for treatment of pelvic floor myalgia. A 2016 retrospective chart review performed at the University of Saskatchewan revealed a reduction in both dyspareunia and pelvic floor muscle spasm with the use of baclofen and diazepam vaginal suppositories.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant pelvic floor dyssynergia and pain during sexual activity.

Exclusion Criteria:

* Decide you do not wish to participate
* Are pregnant
* Have active pelvic inflammatory disease
* Have an active sexually transmitted infection (STI)
* Have a known or suspected cancer of the genital tract
* Have untreated or unevaluated changes in your Pap smear
* Are not currently sexually active
* Have an allergy to either baclofen or valium
* Are unable to complete the necessary study questionnaires

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 46XX women
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale for Pain (VAS-P) scores before and after treatment | 5 months
  The scale ranges from 0 (no pain) to 10 (worst pain ever experienced)

SECONDARY OUTCOMES:
Change in Female Sexual Function Index (FSFI) | 5 months
  Self report measure of female sexual dysfunction
Patient Global Impression of Improvement (PGI-I) | 5 months
  Ranks patients overall feeling about health from 1 (very much better) to 7 (very much worse)
Short form Health Survey (SF-12) | 5 months
  Standardized self assessment tool to measure overall health status

IPD SHARING:
Plan to Share IPD: No
only pooled data will be shared outside of the research team